CLINICAL TRIAL: NCT02369939
Title: Randomized Trial to Evaluate Effects of Deep Regional Hyperthermia in Patients With Anal Carcinoma Treated by Standard Radiochemotherapy
Brief Title: Effects of Deep Regional Hyperthermia in Patients With Anal Carcinoma Treated by Standard Radiochemotherapy
Acronym: HYCAN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYCAN
Record Dates: First submitted 2015-01-07; First posted 2015-02-24 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Anal Carcinoma
Keywords: anal carcinoma; hyperthermia; radiotherapy; chemotherapy; radiochemotherapy
MeSH Terms: conditions — Anus Neoplasms; Hyperthermia | interventions — Radiation; Mitomycin; Fluorouracil; Diathermy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control arm (Active Comparator): Irradiation 1.8Gy/d; T2N0 55.8Gy; T3N0-T4N0 59.4Gy Chemotherapy: Mitomycin C 10mg/m^2/d on d1 and 29; 5-Fluorouracil 1000mg/m^2/d on d1-5, 29-33
  Interventions: Radiation: Irradiation; Drug: Mitomycin C; Drug: 5-Fluorouracil
- Experimental arm (Experimental): Irradiation 1.8Gy/d; T2N0 55.8Gy; T3N0-T4N0 59.4Gy Chemotherapy: Mitomycin C 10mg/m^2/d on d1 and 29; 5-Fluorouracil 1000mg/m^2/d on d1-5, 29-33 Hyperthermia: 6
  Interventions: Radiation: Irradiation; Drug: Mitomycin C; Drug: 5-Fluorouracil; Procedure: Hyperthermia

INTERVENTIONS:
Radiation: Irradiation — Radiotherapy 55,8 Gy - 59,4 Gy
Drug: Mitomycin C — MMC w1, w5
  Other Names: any brand is permitted
Drug: 5-Fluorouracil — 5-FU w1, w5
  Other Names: any brand is permitted
Procedure: Hyperthermia — 6x deep regional hyperthermia
  Other Names: Deep regional hyperthermia
  Arms: Experimental arm

SUMMARY:
Randomized study to investigate the efficacy of deep regional hyperthermia in patients with anal carcinoma treated by standard radiochemotherapy with MMC and 5-FU.

DETAILED DESCRIPTION:
Pat. with anal carcinoma and treated with standard radiochemotherapy with Mitomycin C and 5-FU will in the experimental arm receive deep regional hyperthermia (6x).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven anal squamous cell carcinoma (SCC) (WHO 2004), including anal canal carcinoma (UICC 2002) and anal margin carcinoma (UICC 2002)
* All stages except T1 N0 M0 after local excision (UICC 2002)
* Age ≥ 18 years
* ECOG Status 0-1
* Patients that have understand protocol and signed informed consent form
* Sufficient bone marrow function: WBC ≥ 3,0 x 10^9/l, Platelets ≥ 100 x 10^9/l, Hemoglobin ≥ 10 g/dl
* Sufficient liver function: Bilirubin < 1,5 mg/dl, SGOT, SGPT, alkaline phosphatase, gGT less than 3 times upper limit of normal

Exclusion Criteria:

* Stage T1 N0 M0 after local excision (UICC 2002)
* Uncontrolled, severe cardiac dysfunction (NYHA III/IV)
* Pre-existing uncontrolled cardiac disease, signs of cardiac failure, or rhythm disturbances requiring therapy
* Myocardial infarction within the past 12 months
* Congestive heart failure
* Complete bundle branch block
* New York Heart Association (NYHA) class III or IV heart disease
* Chronic inflammatory disease of the intestine
* Active intractable or uncontrolled infection
* Chronic diarrhea ( > NCI CTC-Grad 1)
* Acute thrombosis
* Collagen vascular disease
* Cardiac pacemaker
* HIV-infection; Patients with hepatitis A or B virus infection, with HPV infection or Patients receiving immune suppressive treatment can be included
* Devices that preclude deep regional hyperthermia (Endoprosthesis, stent in vascular system, acute thrombosis)
* Any metal implants (with exception of non-clustered marker clips)
* Conditions that preclude the application of fractionated pelvic radiotherapy
* Conditions that preclude regular follow-up
* Pregnant or breast feeding women
* Prior pelvic radiotherapy
* Prior chemotherapy
* Drug addiction
* On-treatment participation on other trials
* Prior or concurrent malignancy or leucemia (≤ 5 years prior to enrolment in study) except anal cancer or non-melanoma skin cancer or cervical carcinoma FIGO stage 0-1 if the patient is continuously disease-free
* The presence of increased radiation sensitivity, for example ataxia teleangiectatica, or similar
* Psychological, familial, sociological, or geographical condition that would preclude study compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-12 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Improvement of complete remission | 12 weeks after start of treatment

SECONDARY OUTCOMES:
Colostomy-free survival | 5 years after start of treatment
locoregional relapse-free survival | 5 years after start of treatment
Overall relapse-free survival | 5 years after start of treatment
Overall survival | 5 years after start of treatment
Response rate | 5 years after start of treatment
Rate of acute and late toxicity | 5 years after start of treatment
Quality of life | 5 years after start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Fietkau, Prof. Dr., Study Director — Universitätsklinikum Erlangen, Strahlenklinik
Locations (1):
- Universitaetsklinikum Erlangen, Strahlenklinik, Erlangen, Germany

REFERENCES:
- [Derived] Ott OJ, Schmidt M, Semrau S, Strnad V, Matzel KE, Schneider I, Raptis D, Uter W, Grutzmann R, Fietkau R. Chemoradiotherapy with and without deep regional hyperthermia for squamous cell carcinoma of the anus. Strahlenther Onkol. 2019 Jul;195(7):607-614. doi: 10.1007/s00066-018-1396-x. Epub 2018 Nov 2. PMID 30390114